CLINICAL TRIAL: NCT02825888
Title: Perineural Ultrasound-Guided Axillary Brachial Plexus Block: Influence of Obesity on Block Performance Time, Failure Rate and Incidence of Acute Complications (Observational Study)
Status: Completed | Type: Observational
Sponsor: Dr. Vishal Uppal (Other)
Responsible Party: Sponsor-Investigator, Dr. Vishal Uppal, Fellow/Staff, Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: 103673
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Ultrasound Guided Axillary Brachial Plexus Block
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Non-obese: Body Mass index less than 30 kg/m2
- Obese: Body Mass index more than 30 kg/m2

SUMMARY:
Title of Research Program: Ultrasound Guided Axillary Brachial Plexus Block: Influence of Obesity on Block Failure Rate, Performance Time and Incidence of Acute Complications- A prospective observational cohort study

Background: Axillary brachial plexus (ABP) block is commonly performed as the primary anesthetic technique to provide surgical anesthesia and postoperative analgesia for elbow, forearm and hand surgery. Compared to general anesthesia, ABP blocks have been shown to result in better pain relief, less nausea and vomiting, shortened length of hospital stay, decreased side effects of opioids painkillers and better patient satisfaction. These beneficial effects of ABP blocks are particularly useful for patients who are overweight or obese as this cohort is at a higher risk of experiencing complications from general anesthesia. Traditionally, nerve blocks have been described technically challenging in obese patients. This may not be true now with availability of high-resolution ultrasonography (US). US imaging also allows doctors the ability to visualize the needle "live" to allow for more accurate needle placement. This allows local anesthetic to be placed more precisely resulting in faster onset anesthesia, decreased local anesthetic drug dosages, reduced complications and higher success rate. Ultrasound guidance has not been used for performing ABP block in previous studies in obese patients.

Hypothesis: We hypothesize that the block failure rate is no worse in obese compared to non-obese patients when US guidance is used to perform ABP blocks.

Specific Objectives: The primary objective of this study is to evaluate whether obese patients receiving US guided ABP block as their primary anesthetic modality have a block success rate (defined by a Composite Score ≥ 14 at 30 minutes) worse than their non-obese peers. The secondary objective is to evaluate time parameters around ABP performance, incidence of complications and patient satisfaction.

Methods: This study will be conducted as an observational quasi-experimental multicenter trial at St. Joseph's Health Care (SJHC), London, ON and the Nova Scotia Health Authority (NSHA) Halifax Infirmary (HI) site, Halifax NS. There will be 250 patients taking part in this study. One hundred and fifty patients have already completed the study in Ontario. The duration of the study at the Halifax Infirmary is 10 months. Healthy patients (aged 18-75 years) scheduled to undergo elbow/ forearm/ or hand surgery will be invited to volunteer in this observational study. A study investigator or resident under direction supervision of a study investigator will perform the ABP block. There is NO experimental drug or treatment in this study. Patient demographics including age, sex, arm circumference, height, weight and Body Mass Index will be recorded. Nerve blocks will be performed in a designated area near operating rooms called the block room. US will be used for identification of the nerves supplying the arm and an ABP block will be performed with a total volume of 30 mL of 0.5% ropivacaine according to a standardized procedure. Measurements of sensory and motor blockage will be recorded every 5 minutes for 30 minutes following the ABP block. Block success will be measured and is defined as a score of ≥ 14 on the Composite Score (CS) within 30 minutes of ABP block completion. According to routine care, all patients will receive a phone call from the investigators 24-48 hours after surgery to inquire about complications. The study follows non-inferiority design to show that the success rate in the obese group is not worse than the non-obese when anesthetized. In non-inferiority trials, both intention to treat and per-protocol analysis are recommended; both approaches should support non-inferiority The student's t-test (unpaired, two tailed) will be used for comparison of the means of continuous, normally distributed data or Mann-Whitney U test as appropriate. Categorical data (success rate, complication rate) are to be analyzed using χ2 test or Fisher's exact test, as appropriate. An interim analysis will not be conducted and set at 0.05 for significance and 95% confidence intervals.

Significance/ Importance: This study would provide anesthesiologists additional information to inform their clinical decision-making when dealing with obese patients. To date there are no publications or any registered trials exploring the success rates and technical aspects of ABP blockade in obese patients using US guidance technology for block performance. Therefore, this study is novel and timely for the patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, scheduled to undergo elbow, forearm and hand surgery; Brachial plexus block is offered to patients as a part of planned routine care; American Society of Anesthesiologists' (ASA) status I to III.

Exclusion Criteria:

* Patients with associated significant cardiac and respiratory disease (ASA status IV/V); Any pre-existing medical disorder that would contraindicate an Axillary brachial plexus block i.e. Known hematological disorder or with deranged coagulation parameters, Major organ dysfunction such as hepatic and renal failure, Neuropathy; Allergy to any of the drugs used in the study; Contraindications to brachial plexus block; Cognitive dysfunction that may impair consent or subject ability to complete data collection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects booked for upper limb surgery who have been assessed as potential recipients of PNB during routine preoperative assessment for an expression of interest in study participation.
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Success rate as measured by composite score | 30 minutes after performance of block

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Nova Scotia Health Authority (NSHA) Halifax Infirmary (HI) site, Halifax NS, Halifax
  - St. Joseph's Health Care (SJHC), London-Ontario, London